CLINICAL TRIAL: NCT01376284
Title: Drug Use Investigation for AVOLVE(BPH)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114125
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed dutasteride capsules: Subjects with BPH prescribed dutasteride capsules during study period
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — Collection of safety data

SUMMARY:
The study is designed to investigate the safety and efficacy of dutasteride capsules 0.5 mg collected from the required number of Japanese subjects with benign prostatic hyperplasia (BPH) in order to identify concerns or problems, if any, about the efficacy and safety of its use at post-marketing clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Must be male subjects
* Use dutasteride capsules for the first time

Exclusion Criteria:

* Subjects who is hypersensitivity to dutasteride or 5α reductase inhibitor
* Subjects with severe hepatic function disorder
* Dutasteride capsules shall not be used to female or child

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese male adult subjects with benign prostatic hyperplasia (BPH) who start the treatment with dutasteride capsules
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with BPH treated with dutasteride capsules | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline